CLINICAL TRIAL: NCT02166268
Title: Evaluation of the Efficacy and Safety of AVANZ® Phleum Pratense in Grass Pollen-induced Allergic Rhinitis During Controlled Exposure in an Environmental Challenge Chamber
Acronym: AV-G-03
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AV-G-03; 2013-005130-38 (EudraCT Number)
Record Dates: First submitted 2014-06-11; First posted 2014-06-18 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Grass Pollen Induced Allergic Rhinoconjunctivitis
Keywords: Allergic rhinoconjunctivitis; Allergic rhinitis; Allergy; Grass pollen
MeSH Terms: conditions — Rhinitis, Allergic; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Avanz Phleum pratense (Active Comparator): Avanz Phleum pratense 15,000 SQ+ (standardised quality), suspension for subcutaneous injection.
  Interventions: Drug: AVANZ Phleum pratense 15,000 SQ+
- Placebo (Placebo Comparator): Placebo, suspension for subcutaneous injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AVANZ Phleum pratense 15,000 SQ+
  Arms: Avanz Phleum pratense
Drug: Placebo
  Arms: Placebo

SUMMARY:
The clinical trial will investigate the efficacy of Avanz Phleum pratense in the treatment of rhinitis in an environmental challenge chamber.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Male or female aged 18 to 65 years
* The subject fulfills one of the following criteria:

  * Male
  * Female, infertile
  * Female of child-bearing potential, with a negative pregnancy test
* Moderate-to-severe grass pollen induced rhinoconjunctivitis
* Positive skin prick test response (wheal diameter ≥ 3 mm) to Phleum pratense
* Positive specific Immunoglobulin E (IgE) against Phleum pratense (≥ IgE Class 2; ≥0.70 kilo Unit/L)
* Minimum level of rhinitis symptoms in an grass pollen challenge, defined as a total nasal symptom score of at least 6 (of 12) within the 3-hour grass pollen challenge at performed at the baseline ECC visit
* The subject must be willing and able to comply with the trial protocol

Exclusion Criteria:

* Rhinoconjunctivitis caused by ragweed, mugwort or Alternaria alternate
* Rhinoconjunctivitis caused by animal hair and dander, house dust mites and moulds
* Clinical history of uncontrolled asthma within 3 months prior to screening
* Subjects with reduced lung function forced expiratory volume in 1 second <70% of the predicted value after adequate pharmacologic treatment
* Subjects with asthma requiring treatment with inhaled corticosteroids outside the grass pollen seasons
* Previous treatment with immunotherapy to a grass pollen allergen or a cross reacting allergen within the past 5 years
* Ongoing treatment with any allergen-specific immunotherapy product
* Symptoms of or treatment for upper respiratory tract infection, acute sinusitis, acute otitis media or other relevant infectious process at randomisation and at the baseline challenge
* Clinically relevant nasal polyps
* History of paranasal sinus surgery
* History of surgery of nasal turbinates
* History of anaphylaxis with cardiorespiratory symptoms (immunotherapy, exercise induced, food allergy, drugs or an idiopathic reaction)
* History of recurrent (defined as 2 or more episodes) generalised urticaria during the last 2 years
* History of drug-induced (including immunotherapy) facial angioedema or a family (parents and siblings) history of hereditary angioedema
* Any clinically relevant chronic disease (≥3 months duration) (e.g. cystic fibrosis, malignancy, malabsorption or malnutrition, renal or hepatic abnormality, or any other diseases that in the opinion of the investigator would interfere with the trial evaluations or the safety of the subjects)
* Systemic disease affecting the immune system (e.g. insulin-dependent diabetes, autoimmune disease, immune complex disease, or immune deficiency disease)
* Immunosuppressive treatment (ATC code L04 or L01) within 3 months prior to the screening visit
* Currently treated with tricyclic antidepressants, catecholamine-O
* methyltransferase inhibitors and/or mono amine oxidase inhibitors
* Treatment with antidepressant medication with antihistaminic effect (e.g. doxepin, mianserin)
* Treatment with antipsychotic medications with antihistaminic effect (e.g. chlorpromazine, levomepromazine, clozapine, olanzapine, thioridazine)
* Treatment with anti-IgE drugs (e.g. omalizumab) within 130 days/5 half-lives which ever longest
* Treatment with systemic and/or topical β-blockers
* Use of an investigational drug within 30 days/5 half-lives of the drug, which ever the longest, prior to screening
* History of allergy, hypersensitivity or intolerance to an excipient the investigational drug (except Phleum pratense)
* Being immediate family of the investigator or trial staff, defined as the investigator's/staff's spouse, parent, child, grandparent, or grandchild
* History of alcohol or drug abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2014-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Average total nasal symptom score | After 1-year of treatment
  The Total Nasal Symptom Score consist of 4 symptoms: runny nose, blocked nose, sneezing and itchy nose scored on a scale form 0-3. Measured during the final Environmental challenge chamber (ECC) visit.

SECONDARY OUTCOMES:
Total nasal symptom score collected at the 2nd ECC visit | After 16 weeks of treatment
  The Total Nasal Symptom Score consist of 4 symptoms: runny nose, blocked nose, sneezing and itchy nose scored on a scale form 0-3. Measured during the 2nd ECC visit.
Average Total Symptom Score | Meaured after 16 weeks and 1 year of treatment.
  The total symptom score consist of 4 nasal symptoms and 2 eye symptoms measured on a scale from 0-3. Measured during the 2nd and the final ECC visit
Treatment emergent adverse events | During the 1-year treatment period with Avanz
  Adverse events (AE) will be collected during the trial. AEs will be summaries by treatment group, Medical Dictionary for Regulatory Activities (MedDRA) system organ class, preferred term and broken down by severity, seriousness, action taken, dosing step and outcome. An analysis of local and systemic reactions and AEs leading to discontinuation. An analysis of early and delayed reactions after the treatment will further be performed.

OTHER OUTCOMES:
Average nasal airflow | After 16 weeks and 1-year of treatment
  Average nasal airflow measured via active anterior rhinomanometry measured during the grass pollen challenge in the environmental challenge chamber.
Average nasal secretion | After 16 weeks and 1-year of treatment
  Nasal secretion in pre-weighed handkerchiefs will be collected during each of the ECCs visits.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Hohlfeld, Prof., Principal Investigator — Fraunhofer Institute
Locations (1):
- Fraunhofer Institute, Hanover, Germany